CLINICAL TRIAL: NCT05891769
Title: Evaluation of Patients With Suspected Parathyroid Adenoma and Negative or Equivocal 99mTc Sestamibi SPECT/CT Using 18F Fluorocholine PET/CT
Brief Title: 99mTc Sestamibi SPECT/CT vs 18F Fluorocholine PET/CT
Acronym: 18FCH
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68169
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Parathyroid Adenoma
MeSH Terms: conditions — Parathyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm study enrolling 100 adult participants with suspected parathyroid adenoma and negative or equivocal standard of care 99mTc Sestamibi SPECT/CT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18FCH PET/CT (Experimental): Participant receive 18F Fluorocholine injection and approximately 45-60 minutes later receive a low dose CT scan from skull base to mid thighs, followed by a static PET emission scan over the same area.
  Interventions: Drug: 18Fluorocholine

INTERVENTIONS:
Drug: 18Fluorocholine — 18F Fluorocholine 5 mCi ± 20% administered intravenously.

SUMMARY:
This study proposes the use of a well-established PET isotope, Fluorine-18 (18F), bound to Choline, for a prospective single-center, single-arm study for participants with suspected parathyroid adenoma and negative or equivocal standard of care 99mTc Sestamibi SPECT/CT

ELIGIBILITY:
Inclusion Criteria:

1. Suspected parathyroid adenoma (elevated serum calcium and inappropriately normal or high levels of parathyroid hormone)
2. Negative or equivocal 99mTc Sestamibi SPECT/CT
3. Able to provide written consent
4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 xULN
6. Karnofsky performance status of >50 (or ECOG/WHO equivalent)
7. Women must not be pregnant per the Department of Radiology Policy on Imaging in Potentially Pregnant and Pregnant Women.

Exclusion Criteria:

1. Less than 18 years old at the time of radiotracer administration
2. Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 60 mL/min or serum creatinine >1.5 x ULN
3. QTcF >470 msec on electrocardiogram (ECG) or congenital long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of lesions detected by PET/CT for detecting parathyroid adenomas. | up to 1 hour
  Inclusion criteria suggest recruiting patients with negative or equivocal SPECT/CT, so based on this there will be 0 lesions on SPECT/CT. The goal is to compare/count the number of lesions from PET/CT, if any present versus no lesions with SPECT/CT

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, MD, Study Director — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciappuccini R, Morera J, Pascal P, Rame JP, Heutte N, Aide N, Babin E, Reznik Y, Bardet S. Dual-phase 99mTc sestamibi scintigraphy with neck and thorax SPECT/CT in primary hyperparathyroidism: a single-institution experience. Clin Nucl Med. 2012 Mar;37(3):223-8. doi: 10.1097/RLU.0b013e31823362e5. PMID 22310246
- [Background] Kluijfhout WP, Pasternak JD, Gosnell JE, Shen WT, Duh QY, Vriens MR, de Keizer B, Hope TA, Glastonbury CM, Pampaloni MH, Suh I. 18F Fluorocholine PET/MR Imaging in Patients with Primary Hyperparathyroidism and Inconclusive Conventional Imaging: A Prospective Pilot Study. Radiology. 2017 Aug;284(2):460-467. doi: 10.1148/radiol.2016160768. Epub 2017 Jan 25. PMID 28121522
- [Background] Hope TA, Graves CE, Calais J, Ehman EC, Johnson GB, Thompson D, Aslam M, Duh QY, Gosnell JE, Shen WT, Roman SA, Sosa JA, Kluijfhout WP, Seib CD, Villaneuva-Meyer JE, Pampaloni MH, Suh I. Accuracy of 18F-Fluorocholine PET for the Detection of Parathyroid Adenomas: Prospective Single-Center Study. J Nucl Med. 2021 Nov;62(11):1511-1516. doi: 10.2967/jnumed.120.256735. Epub 2021 Mar 5. PMID 33674400
- [Background] Graves CE, Hope TA, Kim J, Pampaloni MH, Kluijfhout W, Seib CD, Gosnell JE, Shen WT, Roman SA, Sosa JA, Duh QY, Suh I. Superior sensitivity of 18F-fluorocholine: PET localization in primary hyperparathyroidism. Surgery. 2022 Jan;171(1):47-54. doi: 10.1016/j.surg.2021.05.056. Epub 2021 Jul 21. PMID 34301418
- [Background] DeGrado TR, Reiman RE, Price DT, Wang S, Coleman RE. Pharmacokinetics and radiation dosimetry of 18F-fluorocholine. J Nucl Med. 2002 Jan;43(1):92-6. PMID 11801711